CLINICAL TRIAL: NCT04565353
Title: Testing Multiple Behavioral Science Strategies to Increase Flu-Shot Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 843523
Record Dates: First submitted 2020-09-10; First posted 2020-09-25 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Influenza, Human
Keywords: Influenza vaccination; behavioral science interventions; vaccination promotion
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the different arms. Randomization will be stratified by age (65+ vs. 18-64), vaccine receipt in 2019-2020 flu season (yes vs. no/unknown), and study site (Penn Medicine vs. Geisinger).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: As treated participants will receive text messages, there is no scope for blinding. Care providers will not be made aware of subjects' participation in the study, or assigned treatment arms. The study team will only receive data on subjects' assigned arms at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (20):
- Holdout control (No Intervention): Participants will only receive the standard appointment reminders from their providers.
- Default Reservations Opt-Out Condition (Experimental): The day before their scheduled appointment, participants receive a text reading: "A flu shot has been reserved for you to receive at your appointment tomorrow. Reply Y if you want this shot held for you, N if you don't." The text will include a picture of a vial that says "Your Flu Shot" on it.
  Interventions: Behavioral: Flu shot text messages
- Default Reservations Opt-In Condition (Experimental): The day before their scheduled appointment, participants receive a text reading: "Reply Y if you would like to receive a flu shot at your appointment tomorrow, N if not." The text will include a picture of vial with no text on it.
  Interventions: Behavioral: Flu shot text messages
- Intergroup Competition Treatment Condition (Experimental): Three days before their scheduled appointment, participants will receive a text message with information about how much "your region" lagged behind "another region" in flu shot rate last year ("your region" and "another region" will depend on the study site and include realistic flu shot rates based on historical CDC data). Participants will receive a reminder message on the day of the appointment.
  Interventions: Behavioral: Flu shot text messages
- Intergroup Competition Control Condition (Experimental): Three days before their scheduled appointment, participants will receive a text message with information about how much "your region" lagged behind the target flu shot rate of 70% last year ("your region" will depend on the study site and include realistic flu shot rates based on historical CDC data). Participants will receive a reminder message on the day of the appointment.
  Interventions: Behavioral: Flu shot text messages
- Flu Shot for You Symbolic Condition (Experimental): Three days before their scheduled appointment, participants will receive a text message encouraging them to get a flu shot. They will also be told that they have the opportunity to dedicate getting the flu shot to someone by texting back the initials of an individual. Participants will receive a reminder message on the day of the appointment.
  Interventions: Behavioral: Flu shot text messages
- Flu Shot for You Herd Immunity Condition (Experimental): Three days before their scheduled appointment, participants will receive a text message encouraging them to get a flu shot. They will also be told that they have the opportunity of getting the flu shot to protect a vulnerable loved one by texting back the initials of an individual. Participants will receive a reminder message on the day of the appointment.
  Interventions: Behavioral: Flu shot text messages
- Flu Shot for You Control Condition (Experimental): Three days before their scheduled appointment, participants will receive a text message encouraging them to get a flu shot. They will also receive a reminder message on the day of the appointment. They will not receive any further information, nor will they be asked to respond with initials of an individual.
  Interventions: Behavioral: Flu shot text messages
- Prosocial Condition (Experimental): The day before their scheduled appointment, participants will receive a message describing the pro-social benefits of getting a flu shot, and a reminder to ask for their flu shot. The described pro-social benefits will vary whether they emphasize the COVID-19 pandemic (e.g., protecting loved ones from the risk of hospital-acquired COVID-19 infection) or not (e.g., protecting loved ones from serious complications from the flu). Participants will also receive a reminder message on the day of the appointment.
  Interventions: Behavioral: Flu shot text messages
- Self-Oriented Condition (Experimental): The day before their scheduled appointment, participants will receive a message describing the self-oriented benefits of getting a flu shot, and a reminder to ask for their flu shot. The described self-oriented benefits will vary whether they emphasize the COVID-19 pandemic (e.g., protecting oneself from the risk of hospital-acquired COVID-19 infection) or not (e.g., protecting oneself from serious complications from the flu).
  Interventions: Behavioral: Flu shot text messages
- Information Vivid Condition (Experimental): Three days before their scheduled appointment, participants will receive a message inviting them to watch a 2-minute wellness video and answer some related questions, as well as encouragement to get the flu shot. In this condition, the video will contain vivid information about getting the flu. Participants will also receive a reminder message the day before the appointment.
  Interventions: Behavioral: Flu shot text messages
- Information Basic Condition (Experimental): Three days before their scheduled appointment, participants will receive a message inviting them to watch a 2-minute wellness video and answer some related questions, as well as encouragement to get the flu shot. In this condition, the video will contain basic information about getting the flu. Participants will also receive a reminder message the day before the appointment.
  Interventions: Behavioral: Flu shot text messages
- Information Control Condition (Experimental): Three days before their scheduled appointment, participants will receive a message inviting them to watch a 2-minute wellness video and answer some related questions, as well as encouragement to get the flu shot. In this condition, the video will contain information about exercising. Participants will also receive a reminder message the day before the appointment.
  Interventions: Behavioral: Flu shot text messages
- Sharing Humor Condition (Experimental): The day before their scheduled appointment, participants will receive a text message encouraging them to get the flu shot. The message will include a joke about the flu and will encourage participants to share the joke with nurses, doctors, or pharmacists.
  Interventions: Behavioral: Flu shot text messages
- No Humor Condition (Experimental): The day before their scheduled appointment, participants will receive a text message encouraging them to get the flu shot.
  Interventions: Behavioral: Flu shot text messages
- Healthy Habits Easy Health Behavior Condition (Experimental): The day before their scheduled appointment, participants will be asked if they have completed a series of easy health behaviors (e.g., whether they walked 500 feet yesterday, at least two serving of fruits and vegetables in the last week, and slept at least 6 hours the previous night). They will then be encouraged to get a flu shot at their appointment.
  Interventions: Behavioral: Flu shot text messages
- Healthy Habits Difficult Health Behavior Condition (Experimental): The day before their scheduled appointment, participants will be asked if they have completed a series of difficult health behaviors (e.g., whether they walked 3 miles yesterday, ate 4-6 servings of fruits and vegetables yesterday, and slept at least 9 hours the previous night). They will then be encouraged to get a flu shot at their appointment.
  Interventions: Behavioral: Flu shot text messages
- Healthy Habits Control Condition (Experimental): The day before their scheduled appointment, participants will receive a text message encouraging them to get a flu shot.
  Interventions: Behavioral: Flu shot text messages
- Just-In-Time Reminders 24-Hour Condition (Experimental): Seventy-two hours before their appointment, participants will receive a text message alerting them to the availability of the flu vaccine at their upcoming appointment. Participants will be told they'll receive a reminder, which they can opt-out from receiving. The text message reminder will be sent 24 hours before their appointment.
  Interventions: Behavioral: Flu shot text messages
- Just-In-Time Reminders 15-Minute Condition (Experimental): Just-In-Time Reminders 15-Minute Condition: Seventy-two hours before their appointment, participants will receive a text message alerting them to the availability of the flu vaccine at their upcoming appointment. Participants will be told they'll receive a reminder, which they can opt-out from receiving. The text message reminder will be sent 15 minutes before their appointment.
  Interventions: Behavioral: Flu shot text messages

INTERVENTIONS:
Behavioral: Flu shot text messages — Participants will receive text messages per descriptions listed in the arms.
  Arms: Default Reservations Opt-In Condition; Default Reservations Opt-Out Condition; Flu Shot for You Control Condition; Flu Shot for You Herd Immunity Condition; Flu Shot for You Symbolic Condition; Healthy Habits Control Condition; Healthy Habits Difficult Health Behavior Condition; Healthy Habits Easy Health Behavior Condition; Information Basic Condition; Information Control Condition; Information Vivid Condition; Intergroup Competition Control Condition; Intergroup Competition Treatment Condition; Just-In-Time Reminders 15-Minute Condition; Just-In-Time Reminders 24-Hour Condition; No Humor Condition; Prosocial Condition; Self-Oriented Condition; Sharing Humor Condition

SUMMARY:
This research aims to identify which behavioral science strategies are most effective at increasing flu vaccination rates overall and based on patients' individual characteristics. Past behavioral science interventions have shown promise in increasing flu vaccinations. For example, successful interventions have encouraged people to make concrete plans for when they will get a flu vaccination (Milkman et al. 2011), sent automated calls or text messages reminding patients to get a flu vaccination (Cutrona et al. 2018; Regan et al. 2017), or provided financial incentives for getting vaccinated (Nowalk et al. 2010). Although these results are promising, these studies have been conducted in isolation on different populations, which makes it difficult to compare their interventions' effectiveness or to have enough power to reliably detect differing responses to interventions based on individual characteristics.

This research will simultaneously test 19 different SMS interventions to increase flu vaccinations in a "mega-study" and apply machine learning to identify which interventions work best for whom. The interventions are designed by behavioral science experts from the Behavior Change for Good Initiative (BCFG), Penn Medicine Nudge Unit (PMNU), and Geisinger Behavioral Insights Team (BIT). We expect to include at least 80,000 participants.

The specific aims of this research are to identify (1) which behavioral science strategies effectively increase flu vaccination rates overall, and (2) which strategies are most effective for different subgroups (e.g., based on age, gender, race).

ELIGIBILITY:
Penn Medicine and Geisinger patients will be included if they:

Inclusion Criteria:

* Have a cell phone number recorded in a Penn Medicine or Geisinger database
* Have a new or routine primary care appointment during the study recruitment period (not a sick visit)

Exclusion Criteria:

* Have documentation of allergy or adverse event to influenza vaccination in medical records
* Have documentation of already receiving their 2020 influenza vaccination prior to randomization in medical records
* Have opted out of receiving text message appointment reminders
* Have asked not to be contacted for research purposes
* Have an appointment with someone other than their primary care physician
* Have an appointment with someone other than a physician, resident, nurse practitioner, or physician assistant

We will recruit as many patients as possible starting in September 2020. We will stop enrolling participants with appointments scheduled to occur after December 31, 2020 if we have reached 4,000 participants per condition. If we do not have 4,000 participants per condition by December 31, 2020, we will continue enrolling participants until we have reached 4,000 per condition, or until March 31, 2021 (discontinuing enrollment at whichever milestone arrives sooner - 4,000 people enrolled or 3/31/21).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74811 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Geisinger Health, Danville, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Aggregate data and code used for analyses conducted on participants enrolled from September through December is available at https://osf.io/tucjs/?view_only=c491df37a33840abbdedda4e60176f34. This reflects the analyses and data included in this paper: https://www.pnas.org/content/118/20/e2101165118.
  Researchers interested in using individual-level data to replicate our results should contact the Behavior Change for Good Initiative at the University of Pennsylvania (bcfg@wharton.upenn.edu) and must sign a standard medical data nondisclosure agreement to access the data on a protected medical server.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Cutrona SL, Golden JG, Goff SL, Ogarek J, Barton B, Fisher L, Preusse P, Sundaresan D, Garber L, Mazor KM. Improving Rates of Outpatient Influenza Vaccination Through EHR Portal Messages and Interactive Automated Calls: A Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):659-667. doi: 10.1007/s11606-017-4266-9. Epub 2018 Jan 30. PMID 29383550
- [Background] Milkman KL, Beshears J, Choi JJ, Laibson D, Madrian BC. Using implementation intentions prompts to enhance influenza vaccination rates. Proc Natl Acad Sci U S A. 2011 Jun 28;108(26):10415-20. doi: 10.1073/pnas.1103170108. Epub 2011 Jun 13. PMID 21670283
- [Background] Regan AK, Bloomfield L, Peters I, Effler PV. Randomized Controlled Trial of Text Message Reminders for Increasing Influenza Vaccination. Ann Fam Med. 2017 Nov;15(6):507-514. doi: 10.1370/afm.2120. PMID 29133488
- [Background] Nowalk MP, Lin CJ, Toback SL, Rousculp MD, Eby C, Raymund M, Zimmerman RK. Improving influenza vaccination rates in the workplace: a randomized trial. Am J Prev Med. 2010 Mar;38(3):237-46. doi: 10.1016/j.amepre.2009.11.011. Epub 2009 Dec 24. PMID 20036102
- [Derived] Buttenheim A, Milkman KL, Duckworth AL, Gromet DM, Patel M, Chapman G. Effects of Ownership Text Message Wording and Reminders on Receipt of an Influenza Vaccination: A Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e2143388. doi: 10.1001/jamanetworkopen.2021.43388. PMID 35175346

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A small number of patients in each experimental condition did not receive any intervention messages due to technical malfunctions. These patients are excluded from analyses since they were, for all practical purposes, not a part of of our study
Period: Overall Study
Arm/Group | Holdout Control | Default Reservations Opt-Out Condition | Default Reservations Opt-In Condition | Intergroup Competition Treatment Condition | Intergroup Competition Control Condition | Flu Shot for You Symbolic Condition | Flu Shot for You Herd Immunity Condition | Flu Shot for You Control Condition | Prosocial Condition | Self-Oriented Condition | Information Vivid Condition | Information Basic Condition | Information Control Condition | Sharing Humor Condition | No Humor Condition | Healthy Habits Easy Health Behavior Condition | Healthy Habits Difficult Health Behavior Condition | Healthy Habits Control Condition | Just-In-Time Reminders 24-Hour Condition | Just-In-Time Reminders 15-Minute Condition
Started | 3742 | 3737 | 3709 | 3735 | 3758 | 3769 | 3719 | 3732 | 3728 | 3777 | 3672 | 3751 | 3737 | 3714 | 3773 | 3739 | 3776 | 3744 | 3741 | 3758
Completed | 3742 | 3688 | 3670 | 3693 | 3717 | 3716 | 3665 | 3693 | 3662 | 3734 | 3623 | 3710 | 3685 | 3664 | 3736 | 3690 | 3734 | 3696 | 3698 | 3712
Not Completed | 0 | 49 | 39 | 42 | 41 | 53 | 54 | 39 | 66 | 43 | 49 | 41 | 52 | 50 | 37 | 49 | 42 | 48 | 43 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Holdout Control | Default Reservations Opt-Out Condition | Default Reservations Opt-In Condition | Intergroup Competition Treatment Condition | Intergroup Competition Control Condition | Flu Shot for You Symbolic Condition | Flu Shot for You Herd Immunity Condition | Flu Shot for You Control Condition | Prosocial Condition | Self-Oriented Condition | Information Vivid Condition | Information Basic Condition | Information Control Condition | Sharing Humor Condition | No Humor Condition | Healthy Habits Easy Health Behavior Condition | Healthy Habits Difficult Health Behavior Condition | Healthy Habits Control Condition | Just-In-Time Reminders 24-Hour Condition | Just-In-Time Reminders 15-Minute Condition | Total
Number analyzed (Participants) | 3742 | 3737 | 3709 | 3735 | 3758 | 3769 | 3719 | 3732 | 3728 | 3777 | 3672 | 3751 | 3737 | 3714 | 3773 | 3739 | 3776 | 3744 | 3741 | 3758 | 74811
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 24 | 21 | 20 | 31 | 21 | 21 | 15 | 24 | 24 | 22 | 31 | 24 | 14 | 24 | 19 | 16 | 19 | 20 | 28 | 440
  Between 18 and 65 years | 2950 | 2920 | 2921 | 2940 | 2942 | 2941 | 2916 | 2923 | 2932 | 2955 | 2902 | 2948 | 2961 | 2950 | 2942 | 2927 | 2956 | 2932 | 2947 | 2959 | 58764
  >=65 years | 770 | 793 | 767 | 775 | 785 | 807 | 782 | 794 | 772 | 798 | 748 | 772 | 752 | 750 | 807 | 793 | 804 | 793 | 774 | 771 | 15607
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (16.2) | 50.7 (16.4) | 50.5 (16.3) | 50.7 (16.2) | 50.5 (16.2) | 50.9 (16.3) | 50.5 (16.4) | 50.8 (16.6) | 50.9 (16.2) | 50.6 (16.2) | 50.8 (16.1) | 50.8 (16.1) | 50.7 (16.1) | 50.5 (16.2) | 50.9 (16.3) | 51.0 (16.3) | 51.0 (16.0) | 50.7 (16.3) | 50.7 (16.2) | 50.5 (16.0) | 50.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2056 | 2109 | 2079 | 2067 | 2096 | 2097 | 2018 | 2091 | 2083 | 2120 | 2030 | 2107 | 2060 | 2104 | 2098 | 2085 | 2159 | 2120 | 2101 | 2091 | 41771
  Male | 1686 | 1628 | 1630 | 1668 | 1662 | 1672 | 1701 | 1641 | 1645 | 1657 | 1642 | 1644 | 1677 | 1610 | 1675 | 1654 | 1617 | 1624 | 1640 | 1667 | 33040
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race category: Asian | 86 | 82 | 91 | 99 | 86 | 75 | 87 | 88 | 93 | 83 | 90 | 91 | 87 | 88 | 93 | 84 | 80 | 89 | 85 | 77 | 1734
  Race category: Black | 751 | 729 | 736 | 688 | 730 | 717 | 711 | 705 | 719 | 755 | 676 | 667 | 713 | 673 | 741 | 676 | 722 | 714 | 698 | 701 | 14222
  Race category: Hispanic | 187 | 177 | 173 | 168 | 157 | 180 | 156 | 174 | 174 | 177 | 181 | 143 | 177 | 183 | 154 | 160 | 162 | 175 | 145 | 188 | 3391
  Race category: Other | 140 | 114 | 149 | 126 | 134 | 147 | 130 | 116 | 140 | 108 | 139 | 128 | 144 | 131 | 128 | 135 | 113 | 144 | 134 | 138 | 2638
  Race category: White | 2578 | 2635 | 2560 | 2654 | 2651 | 2650 | 2635 | 2649 | 2602 | 2654 | 2586 | 2722 | 2616 | 2639 | 2657 | 2684 | 2699 | 2622 | 2679 | 2654 | 52826

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Flu Shot Receipt at or Before Appointment
Description: Our field experiment will be conducted with Penn Medicine and Geisinger Health patients via SMS messages sent prior to their first primary care appointment during the study period, hereafter referred to as the "target appointment." The key dependent variable is whether participants receive a flu shot at or before their target appointment (as recorded in their electronic health records).
  If participants cancel or do not show up for their target appointment after they have been randomized to a treatment and then schedule a new appointment during the study period, their new primary care appointment becomes the target appointment.
  Participants who have been randomized to a treatment will be counted as not having received a flu shot if they cancel or do not show up for their target appointment and do not schedule a new appointment during the study period.
  Participants who receive a flu shot before they receive the SMS intervention will be excluded from the analyses.
Time Frame: The dependent variable will be assessed during a 4-day period after randomization starting three days prior to the participant's target primary care appointment through the date of the target appointment (including the date of the appointment)
Measure: Count of Participants; unit: Participants
Arm/Group | Holdout Control | Default Reservations Opt-Out Condition | Default Reservations Opt-In Condition | Intergroup Competition Treatment Condition | Intergroup Competition Control Condition | Flu Shot for You Symbolic Condition | Flu Shot for You Herd Immunity Condition | Flu Shot for You Control Condition | Prosocial Condition | Self-Oriented Condition | Information Vivid Condition | Information Basic Condition | Information Control Condition | Sharing Humor Condition | No Humor Condition | Healthy Habits Easy Health Behavior Condition | Healthy Habits Difficult Health Behavior Condition | Healthy Habits Control Condition | Just-In-Time Reminders 24-Hour Condition | Just-In-Time Reminders 15-Minute Condition
Number analyzed (Participants) | 3742 | 3688 | 3670 | 3693 | 3717 | 3716 | 3665 | 3693 | 3662 | 3734 | 3623 | 3710 | 3685 | 3664 | 3736 | 3690 | 3734 | 3696 | 3698 | 3712
Participants | 1113 | 1210 | 1150 | 1163 | 1183 | 1200 | 1192 | 1191 | 1157 | 1224 | 1144 | 1231 | 1171 | 1135 | 1199 | 1181 | 1193 | 1130 | 1240 | 1227

2. Secondary Outcome: Number of Participants With Flu Shot Receipt Before March 31, 2021
Description: The secondary dependent variable is whether participants receive the flu shot at or before their target appointment or at any time after this appointment (by March 31, 2021), as recorded in their electronic health records.
  Participants who receive a flu shot before they receive the SMS intervention will be excluded from the analyses.
Time Frame: Up to 6 months after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Holdout Control | Default Reservations Opt-Out Condition | Default Reservations Opt-In Condition | Intergroup Competition Treatment Condition | Intergroup Competition Control Condition | Flu Shot for You Symbolic Condition | Flu Shot for You Herd Immunity Condition | Flu Shot for You Control Condition | Prosocial Condition | Self-Oriented Condition | Information Vivid Condition | Information Basic Condition | Information Control Condition | Sharing Humor Condition | No Humor Condition | Healthy Habits Easy Health Behavior Condition | Healthy Habits Difficult Health Behavior Condition | Healthy Habits Control Condition | Just-In-Time Reminders 24-Hour Condition | Just-In-Time Reminders 15-Minute Condition
Number analyzed (Participants) | 3742 | 3688 | 3670 | 3693 | 3717 | 3716 | 3665 | 3693 | 3662 | 3734 | 3623 | 3710 | 3685 | 3664 | 3736 | 3690 | 3734 | 3696 | 3698 | 3712
Participants | 1296 | 1391 | 1330 | 1343 | 1338 | 1371 | 1369 | 1370 | 1360 | 1418 | 1316 | 1385 | 1342 | 1310 | 1351 | 1370 | 1360 | 1297 | 1388 | 1388

ADVERSE EVENTS:
Time Frame: 9/20/20 - 3/31/21 -- A period of over six months
Description: This is a minimal risk study, eligible for expedited IRB review in keeping with 45 CFR §46.110. All data is gathered from Electronic Health Records (EHR).
  EHR data will report inputs and outcomes; we will therefore be unable to monitor this data for AE/SAEs. Data will be received at the end of the study and may also be received periodically over the course of the study. Even if we receive data periodically, however, we will not be able to monitor it for AE/SAEs
Arm/Group | Holdout Control | Default Reservations Opt-Out Condition | Default Reservations Opt-In Condition | Intergroup Competition Treatment Condition | Intergroup Competition Control Condition | Flu Shot for You Symbolic Condition | Flu Shot for You Herd Immunity Condition | Flu Shot for You Control Condition | Prosocial Condition | Self-Oriented Condition | Information Vivid Condition | Information Basic Condition | Information Control Condition | Sharing Humor Condition | No Humor Condition | Healthy Habits Easy Health Behavior Condition | Healthy Habits Difficult Health Behavior Condition | Healthy Habits Control Condition | Just-In-Time Reminders 24-Hour Condition | Just-In-Time Reminders 15-Minute Condition
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04565353/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT04565353/SAP_001.pdf